CLINICAL TRIAL: NCT01340911
Title: A Randomized, Placebo-Controlled, Single-Blind, Dose-Escalation, First-Time-in-Human Study to Assess the Safety and Pharmacokinetics of Single and Repeat Doses of SRT3025 in Normal Healthy Volunteers
Brief Title: A Study in Healthy Male Volunteers to Investigate Different Doses of a New Drug for the Treatment of Metabolic Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 115444
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SRT3025

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1A, Cohorts 1-6 (Active Comparator): Approximately 48 healthy male subjects will be enrolled into 6 separate cohorts (8 subjects per cohort). Each Cohort of subjects will be dosed sequentially, approximately one week apart, at escalating doses. Within each cohort, 6 subjects will be randomized to receive a single dose of SRT3025, and 2 will be randomized to receive a single dose of placebo.
  The following are the planned doses for Cohorts 1-6, with Cohort 1 being the lowest dose and Cohort 6 being the highest dose: 50, 150, 500, 1000, 2000, and 3000mg of SRT3025. Dose level may be altered as appropriate during the study based on real time analysis of the safety, tolerability, and /or PK data. Dose adjustment may involve an increase or decrease in dose or dividing the total daily dose allowing for twice-daily dosing. Total daily dosing will not exceed 3000mg.
  Interventions: Drug: SRT3025; Drug: Placebo
- Part 1B, Cohorts 7-8 (Active Comparator): One to two of the doses administered in Part 1A may be selected for administration with food, based on expected changes in SRT3025 exposures with food, as well as safety, tolerability, and PK data from Part 1A. If initiated, the effect of a single dose of SRT3025 with a moderate fat/calorie meal may be initiated concurrently with a cohort in Part 2 of the study. Approximately 6 subjects would be enrolled into each cohort in Part 1B.
  Interventions: Drug: SRT3025
- Part 2A, Cohorts 9-11 (Active Comparator): Approximately 16-24 healthy subjects will be enrolled into 2 to 3 cohorts (8 subjects per cohort) in Part 2A. Within each cohort, 6 subjects will be randomized to receive multiple doses of SRT3025, and 2 will be randomized to receive multiple doses of placebo. The repeat dosing component of the study will be initiated, and doses selected, based on the evaluation of safety, tolerability, and PK data from Part 1A. Subjects in Part 2A will be randomized to receive 14 consecutive days of dosing with SRT3025 or matched-placebo. Subjects in these Cohorts will be dosed sequentially (in the fasted state) approximately two weeks apart.
  Interventions: Drug: SRT3025; Drug: Placebo
- Part 2B, Cohorts 12-13 (Active Comparator): If initiated, the effect of repeat doses of SRT3025 with moderate fat/calorie meals would occur in Part 2B (Cohorts 12 and 13). Each of these cohorts would enroll approximately 6 subjects.
  Interventions: Drug: SRT3025

INTERVENTIONS:
Drug: SRT3025 — SRT3025 will be supplied as hard gelatin capsules containing either 27.4 mg (25 mg SRT3025 free base equivalent) or 274 mg (250 mg SRT3025 free base equivalent) of SRT3025 HCl monohydrate drug substance.
Drug: Placebo — For placebo product, the SRT3025 drug substance will be replaced by Microcrystalline Cellulose (Avicel® PH 105) to match the SRT3025 investigational product.
  Arms: Part 1A, Cohorts 1-6; Part 2A, Cohorts 9-11

SUMMARY:
The main purpose of the study is to see how safe SRT3025 (study drug) is when given at different doses. The study will also investigate how the study drug is taken up, metabolised (chemically broken down), distributed through the body and excreted. A further aim is to look at how taking the study drug after eating might change this process.

DETAILED DESCRIPTION:
SRT3025 is being developed for the treatment of metabolic diseases. This study is the first administration of SRT3025 in humans and seeks to establish the initial safety, tolerability, and pharmacokinetic (PK) profile of SRT3025 (and any metabolites, if analyzed) before proceeding to future Phase 1 studies or Phase 2 patient studies.

This protocol details a Phase 1, randomized, placebo-controlled, single-blind, dose escalation study to determine the safety, tolerability, and PK profile of SRT3025 in healthy male subjects. The study will be conducted in two parts. In Part 1A, 6 Cohorts of subjects will receive single escalating doses of SRT3025. In Part 1B, an additional one to two cohorts may be enrolled to investigate the effect of a moderate fat/calorie meal on single dose PK endpoints. In Part 2A, up to three cohorts may be enrolled to receive 14-day repeat doses of SRT3025 chosen from the Part 1A safety, tolerability, and PK data. In Part 2B, one to two additional cohorts may receive 14-day repeat doses of SRT3025 in combination with a moderate fat/calorie meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the Sirtris Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male between 18 and 55 years of age, inclusive, at the time of signing the informed consent.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods that is permitted in the study. This criterion must be followed from the time of the first dose of study medication until the End of Study Safety Follow-up Visit.
* Body weight ≥50 kilogram (kg) and body mass index (BMI) within the range 18-29.9 kg/m^2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase and bilirubin ≥ 1.5x upper limit normal (ULN) (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin >35%).
* Have an abnormal 12-lead electrocardiogram (ECG) or an ECG with abnormality considered to be clinically significant in the opinion of the Investigator. Specifically, single QTcB > 450 msec; or QTc > 480 msec in subjects with Bundle Branch Block.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the 3 months prior to the first dosing day in the current study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sirtris Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Sirtris Medical Monitor, contraindicates his/her participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma, history of asthma, are experiencing flu-like symptoms, or have had an upper respiratory tract infection within two weeks of screening.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2011-06-03 (Actual); Primary Completion 2011-11-24 (Actual); Study Completion 2011-11-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and incidence of adverse events will be used as a measure of safety and tolerability of a single dose of SRT3025 in healthy male subjects. | 9 days
  Number of participants with adverse events and incidence of adverse events will be used as a measure of safety and tolerability of a single dose of SRT3025 in healthy male subjects.
Number of participants with adverse events and incidence of adverse events will be used as a measure of safety and tolerability of multiple doses of SRT3025 in healthy male subjects. | 21 days
  Number of participants with adverse events and incidence of adverse events will be used as a measure of safety and tolerability of multiple doses of SRT3025 in healthy male subjects.

SECONDARY OUTCOMES:
Plasma levels of SRT3025 will be measured in all subjects that received a single dose of the study drug at fasted and fed states to assess the pharmacokinetics and bioavailability of SRT3025. | 24 hours
  Plasma levels of SRT3025 will be measured in all subjects that received a single dose of the study drug at fasted and fed states to assess the pharmacokinetics and bioavailability of SRT3025.
Plasma levels of SRT3025 will be measured in all subjects that received multiple doses of the study drug at fasted and fed states to assess the pharmacokinetics and bioavailability of SRT3025. | 14 days
  Plasma levels of SRT3025 will be measured in all subjects that received multiple doses of the study drug at fasted and fed states to assess the pharmacokinetics and bioavailability of SRT3025.
SRT3025 metabolite levels in urine and plasma will be measured in all subjects that received a single dose of SRT3025. | 24 hours
  SRT3025 metabolite levels in urine and plasma will be measured in all subjects that received a single dose of SRT3025.
SRT3025 metabolite levels in urine and plasma will be measured in all subjects that received multiple dose of SRT3025. | 15 days
  SRT3025 metabolite levels in urine and plasma will be measured in all subjects that received multiple dose of SRT3025.
Plasma levels of SRT3025 may be compared to the number and types of adverse events experienced by subjects receiving a single dose of SRT3025 to assess any relationship between plasma SRT3025 levels and adverse events. | 9 days
  Plasma levels of SRT3025 may be compared to the number and types of adverse events experienced by subjects receiving a single dose of SRT3025 to assess any relationship between plasma SRT3025 levels and adverse events.
Plasma levels of SRT3025 may be compared to the number and types of adverse events experienced by subjects receiving multiple doses of SRT3025 to assess any relationship between plasma SRT3025 levels and adverse events. | 21 days
  Plasma levels of SRT3025 may be compared to the number and types of adverse events experienced by subjects receiving multiple doses of SRT3025 to assess any relationship between plasma SRT3025 levels and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115444 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115444?search=study&search_terms=115444#rs
- Available data/document: Individual Participant Data Set: 115444 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115444 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115444 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115444 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115444 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115444 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register